CLINICAL TRIAL: NCT06125561
Title: A Study of Periodontal Health and Its Impact on Oral Health-related Quality of Life Among Diabetes Mellitus Patients
Brief Title: Periodontal Health and Its Impact on Oral Health-related Quality of Life Among Diabetes Mellitus Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Pakistan Institute of Medical Sciences (Other Government)
Responsible Party: Principal Investigator, nosheen sarwar, Principle Investigator, Pakistan Institute of Medical Sciences
Other Study IDs: 14112023
Record Dates: First submitted 2023-11-04; First posted 2023-11-09 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Diabetes Mellitus; Periodontal Diseases
MeSH Terms: conditions — Diabetes Mellitus; Periodontal Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Diabetic: Diabetic patients with age ranges 18-60 years. Clinical Examination will be performed by CPTIN probe and questionnaire will be filled by participant's.
  Interventions: Other: Probing depth and Clinical attachment loss
- Non diabetic: Non Diabetic patients with age ranges 18-60 years. Clinical Examination will be performed by CPTIN probe and questionnaire will be filled by participant's.
  Interventions: Other: Probing depth and Clinical attachment loss

INTERVENTIONS:
Other: Probing depth and Clinical attachment loss — CPTIN probe will be used for the clinical examination

SUMMARY:
Periodontal diseases, encompassing a range of inflammatory conditions affecting the supporting structures of the teeth, have long been recognized as a prevalent comorbidity in individuals with diabetes. The severity of periodontal disease is usually documented by research clinicians using clinical parameters such as bleeding on probing (BOP), probing pocket depth (PPD), and clinical.

DETAILED DESCRIPTION:
Oral health plays a pivotal role in the overall well-being and quality of life of individuals. Any condition affecting oral health can have far-reaching consequences for an individual's daily life.Both periodontitis and diabetes have been reported to have negative impacts on aspects of daily living and health-related quality of life. Evidence suggests that oral health problems can adversely affect an individual's physical functioning, social standing and wellbeing, and that it can be difficult to dissociate oral health from general health with regards to impacts on quality of life. Oral health-related quality of life (OHRQoL) can be assessed using the Oral Health Impact Profile-14 (OHIP-14) questionnaire

ELIGIBILITY:
Inclusion Criteria:

* Individuals diagnosed with Diabetes Mellitus for case group, non diabetic patients for control group, Age range between 18 to 60 years, informed consent, Participants with varying degrees of periodontal health

Exclusion Criteria:

* Participants with severe systemic illnesses and habits that may significantly affect oral health or quality of life, Individuals with severe cognitive impairment or psychiatric conditions that hinder their ability to participate and provide informed consent.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The patient presented at dental department of hospital
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2023-11-08 (Estimated); Study Completion 2023-11-08 (Estimated)

PRIMARY OUTCOMES:
oral health-related quality of life | 1 day
  the impact of periodontal health on the oral health-related quality of life

SECONDARY OUTCOMES:
Clinical attachment loss | 1 day
  Probing depth and clinical attachment loss will be measured

CONTACTS AND LOCATIONS:
Locations (1):
- PIMS, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No